CLINICAL TRIAL: NCT01658514
Title: A Randomized, Crossover Study Assessing the Single Dose Pharmacokinetics of Delayed-Release Metformin in Subjects With Renal Dysfunction
Brief Title: Assessing the Behavior of Met DR in Subjects With Kidney Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elcelyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LCRM101
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Met DR (Experimental): One dose of 1000 mg metformin delayed-release
  Interventions: Drug: Met DR
- Met XR (Active Comparator): One dose of 1000 mg metformin extended-release
  Interventions: Drug: Met XR
- Placebo (Placebo Comparator): One dose of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Met DR — metformin delayed-release tablets
  Arms: Met DR
Drug: Met XR — metformin extended-release tablets
  Arms: Met XR
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluated how a single dose of delayed-release metformin (Met DR) behaves in subjects with normal kidney function, mild kidney dysfunction, moderate kidney dysfunction, or severe kidney dysfunction. The safety and tolerability of Met DR was also examined. In addition, this study compared the behavior of a single dose of Met DR with that of extended-release metformin (Met XR) and placebo in subjects with the varying levels of kidney function described above.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 (inclusive) years old at Visit 1 (Screening)
2. Male, or female and met all of the following criteria:

   * Not breastfeeding
   * Negative pregnancy test result at Visit 1 (Screening) (not applicable to postmenopausal or surgically sterile females)
   * Surgically sterile, postmenopausal, or if of childbearing potential, practiced and was willing to continue to practice appropriate birth control during the entire duration of the study
   * Body weight of ≥45 kg
3. Body mass index (BMI) of 18.0 to 40.0 kg/m² (inclusive) at Visit 1 (Screening)
4. Had type 2 diabetes mellitus and an HbA1c ≤10.0%
5. Had a physical examination with no clinically significant abnormalities as judged by the investigator
6. Estimated glomerular filtration rate (eGFR) ≥15 mL/min/1.73 m² based on the Modification of Diet in Renal Disease (MDRD) equation
7. Ability to understand and willingness to adhere to protocol requirements

Exclusion Criteria:

1. Had End Stage Renal Disease requiring dialysis or severe renal dysfunction with eGFR <15 mL/min/1.73 m²
2. Was on dialysis or had been on dialysis within 12 months of Visit 1 (Screening)
3. Had received or planned to receive any iodinated contrast dye within 1 week prior to Visit 1 (Screening) or after study medication administration
4. Was taking or had taken within 1 week of Visit 1 cationic drugs that are eliminated by renal tubular secretion (e.g., amiloride, digoxin, morphine, procainamide, quinidine, quinine, ranitidine, triamterene, trimethoprim, and vancomycin)
5. Had a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the investigator, including but not limited to the following conditions:

   * Hepatic disease
   * Gastrointestinal disease
   * Endocrine disorder (type 2 diabetes mellitus was allowed)
   * Cardiovascular disease
   * Central nervous system diseases
   * Psychiatric or neurological disorders
   * Organ transplantation
   * Chronic or acute infection
   * Orthostatic hypotension, fainting spells or blackouts
   * Allergy or hypersensitivity
6. Had any chronic disease requiring medication that had been adjusted in the past 14 days (subjects could take acute intermittent over-the-counter medications such as Tylenol, if needed)
7. Had major surgery of any kind within 6 months of Visit 1 (Screening)
8. Had a clinically significant finding of an electrocardiogram (ECG) as assessed by the investigator at Visit 1 (Screening)
9. Had clinical laboratory test (clinical chemistry, hematology, or urinalysis) abnormalities, other than those related to diabetes or renal disease and other stable diseases, judged by the investigator to be clinically significant at Visit 1 (Screening)
10. Had a hemoglobin result <8 g/dL or a level indicating severe anemia of renal origin
11. Had a physical, psychological, or historical finding that, in the investigator's opinion, would make the subject unsuitable for the study
12. Had received Byetta® or short-acting insulin within 3 days of Visit 1 (Screening)
13. Had received metformin within 4 weeks of Visit 1 (Screening)
14. Had any drug treatment that affects gastrointestinal motility or gastric pH (prescription or over-the-counter), including any antacids or medications such as Rolaids or Pepcid, within 2 days of Visit 2
15. Abused drugs or alcohol or had a history of abuse that in the investigator's opinion would cause the individual to be noncompliant with study procedures
16. Smoked more than 10 cigarettes, 3 cigars, or 3 pipes per day
17. Had donated blood within 2 months of Visit 1 (Screening) or was planning to donate blood during the study
18. Had received any investigational drug within one month (or seven half-lives of the investigational drug, whichever was greater) of Visit 1 (Screening)
19. Had known allergies or hypersensitivity to any component of study treatment
20. Was employed by Elcelyx Therapeutics, Inc (that is an employee, temporary contract worker, or designee of the company)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Canas, MD, Principal Investigator — Prism Research; Kenneth Lasseter, MD, Principal Investigator — Clinical Pharmacology of Miami, Inc; Alexander White, MD, Principal Investigator — Progressive Medical Research; Harold Bays, MD, Principal Investigator — Louisville Metabolic and Atherosclerosis Research Center; Craig Curtis, MD, Principal Investigator — Compass Research; Prabir Roy-Chaudhury, Principal Investigator — Cincinnati Veterans Affairs Medical Center Department of Internal Medicine; Sunder Mudaliar, Principal Investigator — San Diego Veterans Healthcare System; Nelson Kopyt, Principal Investigator — Northeast Clinical Research Center

REFERENCES:
- [Result] Bakris GL, Mudaliar, S, Kim T, Burns C, Skare S, Baron A, Fineman M. Effects of New Metformin Formulation in Stage 3 and 4 CKD: A Pilot Study. J Am Soc Nephrol. 2014; 25:549A.
- [Result] DeFronzo R, Fleming GA, Chen K, Bicsak TA. Metformin-associated lactic acidosis: Current perspectives on causes and risk. Metabolism. 2016 Feb;65(2):20-9. doi: 10.1016/j.metabol.2015.10.014. Epub 2015 Oct 9. PMID 26773926

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence ABC; Sequence CAB; Sequence BCA: A = 1 dose of 1000 mg Met XR B = 1 dose of 1000 mg Met DR C = 1 dose of placebo
  each treatment was separated by a wash out period of 2 to 10 days
Period: Overall Study
Arm/Group | Sequence ABC | Sequence CAB | Sequence BCA
Started | 14 | 11 | 14
Completed Treatment A | 14 | 11 | 12
Completed Treatment B | 13 | 11 | 14
Completed Treatment C | 13 | 11 | 12
Started - Normal RF Cohort Only | 3 | 2 | 3
Completed - Normal RF Cohort Only | 3 | 2 | 3
Started - Mild RI Cohort Only | 4 | 3 | 4
Completed - Mild RI Cohort Only | 4 | 3 | 4
Started - Moderate RI Cohort Only | 4 | 4 | 4
Completed - Moderate RI Cohort Only | 3 | 4 | 2
Started - Severe RI Cohort Only | 3 | 2 | 3
Completed - Severe RI Cohort Only | 3 | 2 | 3
Completed | 13 | 11 | 12
Not Completed | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Population - All subjects were to receive all interventions and are distributed in this module according to their renal function cohort to inform PK analyses comparing these populations
Groups:
- Normal: Normal Renal Function = eGFR ≥90 mL/min/1.73 m²
- Mild RI: Mild Renal Impairment = eGFR ≥60 to <90 mL/min/1.73 m²
- Moderate RI: Moderate Renal Impairment = eGFR ≥30 to <60 mL/min/1.73 m²
- Severe RI: Severe Renal Impairment = eGFR ≥15 to <30 mL/min/1.73 m²
- Total: Total of all reporting groups
Arm/Group | Normal | Mild RI | Moderate RI | Severe RI | Total
Number analyzed (Participants) | 8 | 11 | 12 | 8 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.01) | 60.8 (6.62) | 72.6 (3.90) | 70.5 (5.50) | 65.1 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 0 | 1 | 7
  Male | 6 | 7 | 12 | 7 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 8 | 10 | 10 | 8 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 5 | 2 | 4 | 12
  White | 7 | 6 | 10 | 3 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: kg] | 94.9 (18.02) | 94.9 (12.06) | 94.2 (14.96) | 99.8 (10.69) | 95.7 (13.73)
BMI [Mean (Standard Deviation); unit: kg/m²] | 32.8 (3.81) | 31.8 (3.79) | 30.4 (3.33) | 33.3 (4.09) | 31.9 (3.75)

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-t) of Plasma Metformin
Description: AUC (0-t) = Area under the curve from the time of dosing (0 h) to the time of the last quantifiable concentration following dose administration
Time Frame: from the time of dosing (0 h) to 72 hours postdose
Population: PK Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: ng*h/mL
Arm/Group | Met DR | Met XR
Number analyzed (Participants) | 34 | 34
ng*h/mL
  Normal (N = 8) | 5362 (943) | 10411 (1831)
  Mild RI (N = 10) | 8705 (1368) | 11788 (1853)
  Moderate RI (N = 9) | 11477 (1915) | 20240 (3377)
  Severe RI (N = 7) | 22893 (4307) | 43683 (8218)
Statistical Analysis 1: Comparison: Met DR vs Met XR; For the Normal Renal Function Cohort. Met XR is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0011, ANOVA — p-values <0.10 are considered statistically significant; Included treatment, renal group, sequence, period and treatment*renal group as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 51.5, 90% CI 2-sided [37.77 to 70.23]
Statistical Analysis 2: Comparison: Met DR vs Met XR; For the Mild RI Renal Function Cohort. Met XR is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0733, ANOVA — p-values <0.10 are considered statistically significant; [statistical method as in outcome 1, analysis 1]; % Ratio of LS Means = 73.8, 90% CI 2-sided [55.97 to 97.43]
Statistical Analysis 3: Comparison: Met DR vs Met XR; For the Moderate RI Renal Function Cohort. Met XR is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0028, ANOVA — p-values <0.10 are considered statistically significant; [statistical method as in outcome 1, analysis 1]; % Ratio of LS Means = 56.7, 90% CI 2-sided [42.25 to 76.10]
Statistical Analysis 4: Comparison: Met DR vs Met XR; For the Severe RI Cohort. Met XR is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0025, ANOVA — p-values <0.10 are considered statistically significant; [statistical method as in outcome 1, analysis 1]; % Ratio of LS Means = 52.4, 90% CI 2-sided [37.61 to 73.02]

2. Primary Outcome: Cmax of Plasma Metformin
Description: Cmax = Maximum concentration from the time of dosing (0 h) to the time of the last quantifiable metformin concentration following dose administration
Time Frame: from the time of dosing (0 h) to 72 hours postdose
Population: PK Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Met DR | Met XR
Number analyzed (Participants) | 34 | 34
ng/mL
  Normal (N = 8) | 969 (153) | 1479 (234)
  Mild RI (N = 10) | 1036 (147) | 1340 (189)
  Moderate RI (N = 9) | 925 (139) | 1634 (245)
  Severe RI (N = 7) | 1414 (239) | 2590 (438)
Statistical Analysis 1: Comparison: Met DR vs Met XR; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0474, ANOVA — p-values <0.10 are considered statistically significant; [statistical method as in outcome 1, analysis 1]; % Ratio of LS Means = 65.5, 90% CI 2-sided [46.32 to 92.68]
Statistical Analysis 2: Comparison: Met DR vs Met XR; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1691, ANOVA — p-values <0.10 are considered statistically significant; [statistical method as in outcome 1, analysis 1]; % Ratio of LS Means = 77.3, 90% CI 2-sided [56.72 to 105.41]
Statistical Analysis 3: Comparison: Met DR vs Met XR; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0064, ANOVA — p-values <0.10 are considered statistically significant; [statistical method as in outcome 1, analysis 1]; % Ratio of LS Means = 56.6, 90% CI 2-sided [40.73 to 78.63]
Statistical Analysis 4: Comparison: Met DR vs Met XR; For the Severe RI Renal Function Cohort. Met XR is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0097, ANOVA — p-values <0.10 are considered statistically significant; [statistical method as in outcome 1, analysis 1]; % Ratio of LS Means = 54.6, 90% CI 2-sided [37.68 to 79.11]

3. Primary Outcome: Correlation of Placebo-adjusted Change From Pre-dose Value in Lactate Versus Metformin Concentration
Description: To determine the exposure-response relationship of metformin and plasma lactate concentrations
Time Frame: from the time of dosing (0 h) to 24 hours postdose
Population: PD Evaluable Population
Measure: Number; unit: R²
Arm/Group | Met DR | Met XR
Number analyzed (Participants) | 34 | 34
R² | 0.000011129 | 0.069527
Statistical Analysis 1: Comparison: Met DR; Test type: Superiority or Other; p = 0.9444, Pearson Correlation — R² for Placebo-adjusted Change from Pre-dose Value in Lactate Versus Metformin Concentration
Statistical Analysis 2: Comparison: Met XR; Test type: Superiority or Other; p < 0.0001, Pearson Correlation — R² for placebo-adjusted change from pre-dose value in lactate versus metformin concentration

ADVERSE EVENTS:
Time Frame: Approximately 19 to 76 days depending on the number of days before the start of Visits 2 and 3 and the number of washout days between the treatment visits.
Arm/Group | Placebo | Met DR | Met XR
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 4/36 | 12/38 | 11/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Met DR (N=38) | Met XR (N=37)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 4
Vessel Puncture Site Haemorrhage (General disorders) | 0 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Infusion Site Haemorrhage (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Vessel Puncture Site Pain (General disorders) | 0 | 0 | 1
Vessel Puncture Site Reaction (General disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study may be published by INSTITUTE, however the publication shall not disclose any SPONSOR Confidential Information, the INSTITUTE shall send the SPONSOR a copy of any such proposed publication 90 days prior to submission for publication, the INSTITUTE, on request of the SPONSOR, shall delete any SPONSOR Confidential Information in the proposed publication, and the INSTITUTE shall, on the SPONSOR's request, delay submission while the SPONSOR files applications for patents.